CLINICAL TRIAL: NCT01341496
Title: Epigenetically-Modified Autologous Tumor Cell Vaccs and ISCOMATRIX(TM) Adjuvant With Metronomic Oral Cyclophosphamide and Celecoxib in Pts Undergoing Resection of Sarcomas, Melanomas, Germ Cell Tumors, or Epithelial Malignancies Metastatic to Lungs, Pleura or Mediastinum
Brief Title: Tumor Cell Vaccines and ISCOMATRIX With Chemotherapy After Tumor Removal
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 110148; 11-C-0148
Record Dates: First submitted 2011-04-22; First posted 2011-04-25 (Estimated); Last update posted 2018-07-05 (Actual); Status verified 2016-07-21

CONDITIONS: Sarcoma; Melanoma; Epithelial Malignancies; Pleural Malignancy
Keywords: Metastatic Cancer; Cancer Vaccine; Immunotherapy; Chest Metastases; Sarcoma; Melanoma
MeSH Terms: conditions — Sarcoma; Melanoma; Neoplasm Metastasis | interventions — Cyclophosphamide; Celecoxib

ARMS (1):
- 1 (Experimental): autologous tumor vaccine plus chemotherapy
  Interventions: Biological: Epigenetically Modified Autologous Tumor; Drug: Cyclophosphamide; Drug: Celecoxib

INTERVENTIONS:
Biological: Epigenetically Modified Autologous Tumor — 5x 10^7 autologous tumor cells emulsified in 0.5 mL ISCOMATRIX adjuvant will be administered IM every 4 weeks for 6 months
Drug: Cyclophosphamide — 50 mg PO BID for 7 days prior to the first dose of vaccine and then on days 8 through 14, and 22 through 28 of each 4 week treatment cycle
Drug: Celecoxib — 400 mg PO BID for 7 days prior to the first dose of vaccine and then on days 1 through 28 of each 4 week vaccine cycle.

SUMMARY:
Background:

- A tumor cell vaccine is an experimental cancer treatment. Cancer cells are collected from a patient and then used to develop a vaccine. The vaccine will produce an immune system response to help destroy other cancer cells in the body. Researchers are studying ways to improve these tumor cell vaccines. One way is to add an adjuvant. An adjuvant is a substance that brings about a stronger immune system response. ISCOMATRIX is an adjuvant that has been used safely in other clinical studies. But it has not been studied with certain tumor cell vaccines. Researchers want to find out whether a tumor cell vaccine with ISCOMATRIX, given along with cancer drug treatment, is a safe and effective way to slow or prevent tumor growth after tumor removal surgery.

Objectives:

- To assess the safety and effectiveness of tumor cell vaccines given with ISCOMATRIX and drug therapy after tumor removal surgery.

Eligibility:

- People at least 18 years of age who have had tumor cell vaccines developed from cells taken from surgically removed tumors.

Design:

* Patients will be screened with a physical examination, medical history, blood and urine tests, and imaging studies.
* Patients will be treated with cyclophosphamide (once daily) and celecoxib (twice daily) for 7 days before the first vaccine dose.
* Patients will receive the tumor cell vaccine once a month for 6 months. They will continue to receive drug therapy throughout the vaccine treatment. Patients will be monitored with regular blood tests and imaging studies.
* After the first 6 months, patients who have an immune response to the vaccine will continue treatment with the vaccine and chemotherapy. They will also have regular blood tests and imaging studies. They will have this treatment for up to 24 months from the first vaccination or until they no longer have an immune response.
* Participants will have followup visits for up to 5 years after the first vaccination, or until the tumor returns.

DETAILED DESCRIPTION:
Background:

Cancer-testis (CT) antigens (CTAs) have emerged as attractive targets for cancer immunotherapy. Whereas cancers of various histologies exhibit CTA expression, primary or vaccine-induced immune responses to these antigens appear uncommon in patients with these malignancies, possibly due to low-level, heterogeneous antigen expression, and inadequate vaccination strategies. Because numerous CT antigens can be induced in tumor cells by DNA demethylating agents and HDAC inhibitors, it is conceivable that vaccination of cancer patients with autologous tumor cells exposed to chromatin remodeling agents will enhance anti-tumor immunity in these individuals. In order to examine this issue, patients undergoing complete resection of sarcomas, melanomas, germ cell tumors and epithelial malignancies metastatic to the lungs, pleura or mediastinum will be vaccinated with autologous tumor cells exposed ex-vivo to decitabine and radiation following completion of appropriate combined modality therapy. Vaccines will be administered in conjunction with ISCOMATRIX adjuvant as well as metronomic oral cyclophosphamide (50 mg PO BID x 7d q 14d), and celecoxib (400 mg PO BID). Serologic responses to a variety of recombinant CTAs as well as delayed type hypersensitivity to autologous epigenetically modified tumor cells will be assessed before and after vaccination.

Primary Objective:

-To assess the safety of an epigenetically modified autologous tumor cell vaccine administered with ISCOMATRIX adjuvant in combination with metronomic oral cyclophosphamide and celecoxib in patients undergoing thoracic metastasectomy.

Eligibility:

* Patients with histologically or cytologically proven or clinically evident sarcoma, melanoma, or epithelial malignancies metastatic to lungs, pleura or mediastinum who can be rendered no evidence of disease (NED) by metastasectomy.
* Patients must be 18 years or older with an ECOG performance status of 0 2, without evidence of unstable or decompensated myocardial disease. Patients must have adequate pulmonary reserve evidenced by FEV1 and DLCO equal to or greater than 30% predicted; pCO2 less than 50 mm Hg and pO2 greater than 60 mm Hg on room air ABG; and be on no immunosuppressive medications except inhaled corticosteroids at the time vaccination commences.
* Patients must have a platelet count greater than 100,000, an ANC equal to or greater than 1500 without transfusion or cytokine support, a normal PT, and adequate hepatic function as evidenced by a total bilirubin of <1.5 x upper limits of normal. Serum creatinine less than or equal to 1.6 mg/ml or the creatinine clearance must be greater than 70 ml/min/1.73m(2) at the time vaccination commences.

Design:

* Patients will undergo thoracic metastasectomy using standard of practice guidelines.
* Portions of the resected tumors will be transferred to the Thoracic Oncology Laboratory. Cells will be processed to establish a cancer cell line.
* Following recovery from surgery and appropriate adjuvant chemotherapy and/or radiation, patients will be vaccinated with epigenetically-modified autologous tumor cells periodically over 6 months in conjunction with metronomic oral cyclophosphamide and celecoxib.
* Systemic toxicities and delayed type hypersensitivity responses to autologous tumor cells and serologic responses to a variety of CT antigens will be assessed before and after vaccination.
* Patients will be followed with routine staging scans until disease recurrence.
* As the exact set of comparisons and analyses to be performed will be determined following completion of the trial, and will be based on limited numbers of patients, the analyses will be considered exploratory and hypothesis generating rather than definitive.
* Approximately 80 patients will be accrued to this trial in order to obtain up to 20 evaluable patients.

ELIGIBILITY:
* INCLUSION CRITERIA:

INCLUSION CRITERIA PRIOR TO SURGERY (SCREENING CONSENT):

1. Patients with clinically evident or histologically proven sarcomas, melanomas, germ cell tumors, or epithelial malignancies metastatic to the lungs, mediastinum, or pleura who can be rendered no evidence of active disease (NED) following standard surgical therapy. Note: Patients with active disease outside the thorax may be eligible for the study once the extrathoracic disease is definitively treated by local modalities such as radiation, surgery, or radiofrequency ablation.
2. Patients must have received or refused first line standard systemic therapy for their metastases.
3. Patients with no more than 3 intracranial metastases, which have been definitively treated by surgery or radiation therapy may be eligible for study provided there is no evidence of active disease for at least 2 months.
4. Patients must have an ECOG performance status of 0 2.
5. Patients must be 18 years of age or older due to the unknown effects of immunologic responses to germ cell-restricted gene products during childhood and adolescent development.
6. Seronegative for HIV antibody. Note: The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune competence and thus may be less responsive to the experimental treatment.
7. Seronegative for active hepatitis B, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by RT-PCR and be HCV RNA negative.
8. Patients must be aware of the neoplastic nature of their illnesses, the experimental nature of the therapy, alternative treatments, potential benefits, and risks.
9. Patients must be willing to sign an informed consent and undergo resection of their malignancies at the NCI, to ensure vaccine development.

INCLUSION CRITERIA FOR TREATMENT PHASE OF PROTOCOL (Standard Consent):

1. Patients must have signed the Screening Consent.
2. NCI Laboratory of Pathology confirmation of diagnosis of sarcomas, melanomas, germ cell tumors, or epithelial malignancies metastatic to the lungs, mediastinum, or pleura must have been obtained
3. Patients who were initially rendered NED by surgical resection must remain NED at the time of treatment.
4. Patients with no more than 3 intracranial metastases, which have been definitively treated by surgery or radiation therapy may be eligible for the study, provided there is no evidence of active disease for at least 2 months and no requirement for anticonvulsant therapy or steroids following treatment.
5. Patients must have an ECOG performance status of 0 2.
6. Patients must have evidence of adequate bone marrow reserve, hepatic and renal function as evidenced by the following laboratory parameters:

   Absolute neutrophil count greater than 1500/mm3

   Platelet count greater than 100,000/mm3

   Hemoglobin greater than 8g/dl ( patients may receive transfusions to meet this parameter

   PT within 2 seconds of the ULN

   Total bilirubin <1.5 x upper limits of normal

   Serum creatin ine less than or equal to 1.6 mg/ml or the creatinine clearance must be greater than 70 ml/min/1.73m2.
7. Seronegative for HIV antibody. Note: The experimental treatment being evaluated in this protocol depends on an intact immune system.

   Patients who are HIV seropositive can have decreased immune competence and thus may be less responsive to the experimental treatment.
8. Seronegative for active hepatitis B, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by RT-PCR and be HCV RNA negative.
9. Patients must be willing to practice birth control during and for four months following treatment.
10. Patients must be willing to sign the standard informed consent.

EXCLUSION CRITERIA

1. Patients requiring corticosteroids (other than inhaled) will be excluded.
2. Patients with life expectancy less than 12 months will be excluded.
3. Patients receiving warfarin anticoagulation, who cannot be transferred to other agents such as enoxaparin or dabigatran, and for whom anticoagulants cannot be held for up to 24 hours will be excluded.
4. Patients with uncontrolled hypertension (>160/95), unstable coronary disease evidenced by uncontrolled arrhythmias, unstable angina,decompensated CHF (>NYHA Class II), or myocardial infarctionwithin 6 months of study will be excluded.
5. Patients with other cardiac diseases may be excluded at the discretion of the PI following consultation with Cardiology consultants.
6. Patients with any of the following pulmonary function abnormalities will be excluded: FEV, < 30% predicted; DLCO < 30% predicted (post-bronchodilator); pO2 < 60% or pCO2 (Bullet) 50 on room air arterial blood gas.
7. Pregnant and/or lactating women will be excluded due to the unknown, potentially harmful effects of immune response to CT-X antigens and stem cell proteins that may be expressed in placenta, fetus, and neonates.
8. Patients with active infections, including HIV, will be excluded, due to unknown effects of the vaccine on lymphoid precursors.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-04-18; Primary Completion 2016-05-12 (Actual); Study Completion 2016-07-21 (Actual)

PRIMARY OUTCOMES:
tabulation and grade of observed patient toxicities attributed to the vaccine, and report of the fractions of patients who encounter these toxicities at the various grades | 5 years

SECONDARY OUTCOMES:
Determine if 5 or greater of the first 20 vaccinated patients undergoing thoracic metastasectomy have successful tumor cell line development | 2-3 years
Number and characteristics of immunologic responses to a panel of CT antigens in vaccinated patients | 7 years

CONTACTS AND LOCATIONS:
Overall Officials: David S Schrump, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Quiros RM, Scott WJ. Surgical treatment of metastatic disease to the lung. Semin Oncol. 2008 Apr;35(2):134-46. doi: 10.1053/j.seminoncol.2007.12.010. PMID 18396199
- [Background] ALEXANDER J, HAIGHT C. Pulmonary resection for solitary metastatic sarcomas and carcinomas. Surg Gynecol Obstet. 1947 Aug;85(2):129-46. No abstract available. PMID 20253078
- [Background] Klapper JA, Davis JL, Ripley RT, Smith FO, Nguyen DM, Kwong KF, Mercedes L, Kemp CD, Mathur A, White DE, Dudley ME, Wunderlich JR, Rosenberg SA, Schrump DS. Thoracic metastasectomy for adoptive immunotherapy of melanoma: a single-institution experience. J Thorac Cardiovasc Surg. 2010 Dec;140(6):1276-82. doi: 10.1016/j.jtcvs.2010.05.020. Epub 2010 Jul 2. PMID 20584535